CLINICAL TRIAL: NCT02312700
Title: Development of an Interactive Empowerment Tool in Support of Patient Empowerment.
Brief Title: An Interactive Empowerment Tool for Breast Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Alessandra Gorini, Researcher, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 270089
Record Dates: First submitted 2014-11-28; First posted 2014-12-09 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Breast Cancer; Empowerment
Keywords: empowerment; communication; shared decision making
MeSH Terms: conditions — Breast Neoplasms; Empowerment; Communication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interactive empowerment (IEm) group (Experimental): Intervention: Patients fill in the questionnaire online and their profile (obtained from their answers) is immediately sent to the physician
  Interventions: Behavioral: Interactive empowerment tool
- Control (Sham Comparator): Intervention: Patients fill in the questionnaire online, but their profile (obtained from their answers) is not sent to the physician
  Interventions: Behavioral: Interactive empowerment tool

INTERVENTIONS:
Behavioral: Interactive empowerment tool

SUMMARY:
The study is aimed to verify the effect of an online interactive tool on patient empowerment. The tool is based on a validated psychological questionnaire administrated to breast cancer patients before their first encounter with physician.

DETAILED DESCRIPTION:
The study is intended to develop an IEm (Interactive Empowerment) tool aimed at enhancing physician-patient experience by providing physicians a personalized patient's profile, accompanied by a list of recommendations to suggest him how to interact with that specific patient on the basis of his/her personal profile. Developed in the framework of the FP7 project "P-Medicine", the IEm tool uses the ALGA-BC questionnaire, a recent validated instrument specifically developed to perform a brief evaluation of the breast cancer patients' psychological status, to provide the physician a patient's profile based on 8 factors. As soon as the questionnaire has been completed, the patient's answers are automatically elaborated and sent to the physician's computer. Provided to the physicians at the very beginning of the visit, such information is supposed to be crucial for them to find a tailored way to communicate with the patient. Moreover, in order to help physicians to correctly interpret the patient's score, any time the scores are out of a certain range (normal values) they will receive a recommendation that helps them to find the best way to interact with the patient. Supposing that the patient empowerment can be reached through the improved patient's participation in the clinical process, we argue that a more effective and personalized interaction between patient and physician may have a key role in promoting it.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is aged 18 to 74 years at randomisation.
2. The patient has been diagnosed as having a primary breast cancer requiring a radical surgery
3. The patient is able to understand the Informed Consent Form, and understand study procedures.
4. The patient has signed the Informed Consent Form.

Exclusion Criteria:

1. The patient has a recurrent breast cancer diagnosis
2. The patient has an overt psychiatric illness that would interfere with the measurement of the psychological variables included in the questionnaire
3. Inability to freely consent to take part in the study
4. Inability to understand the study materials.
5. Current participation in another clinical trial relating to the breast cancer treatment
6. Any condition that, in the researcher's opinion, compromises the subject's ability to meet protocol requirements or to complete the study.

Ages: 18 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Improvements in the Patient Empowerment Score | Up to 30 min after the visit
  Patient empowerment score will be measured in the experimental versus the control group by mean of patients' comprehension level relatively to the information doctors provided to them.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Munzono, MD, Principal Investigator — European Institute of Oncology

REFERENCES:
- [Background] Kondylakis H, Kazantzaki E, Koumakis L, Genitsaridi I, Marias K, Gorini A, Mazzocco K, Pravettoni G, Burke D, McVie G, Tsiknakis M. Development of interactive empowerment services in support of personalised medicine. Ecancermedicalscience. 2014 Feb 11;8:400. doi: 10.3332/ecancer.2014.400. eCollection 2014. PMID 24567757
- See also: Web page of the European project in which the present trial is included — http://www.p-medicine.eu